CLINICAL TRIAL: NCT00811486
Title: Body Volume Regulation in Pulmonary Arterial Hypertension With Right Ventricular Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 1 patient recruited, and he withdrew
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-1022
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Right Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Spironolactone; conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Group II
- Spironolactone and conivaptan (Experimental): Group I
  Interventions: Drug: Spironolactone and conivaptan

INTERVENTIONS:
Drug: Spironolactone and conivaptan — Tablet, 50 mg to 200 mg, daily, orally 20 mg intravenously one time over 30 minutes
  Arms: Spironolactone and conivaptan

SUMMARY:
Secondary hyperaldosteronism and the non-osmotic release of arginine vasopressin (AVP) are the major factors in sodium and water retention in pulmonary arterial hypertension with right ventricular failure. Natriuretic doses of mineralocorticoid antagonist and aquaretic doses of V2 receptor antagonist will attenuate the sodium and water retention respectively, and be associated with clinical improvement.

DETAILED DESCRIPTION:
Much has been learned about the pathophysiological state that underlies the development of increased total body volume and edema in left ventricular failure. Very little, however, is known about the mechanism underlying systemic hypervolemia in patients with isolated right ventricular dysfunction. Patients with pulmonary arterial hypertension (PAH) represent a model of isolated right ventricular dysfunction in which these mechanisms may be elucidated. Aldosterone has now been shown to have many properties that are likely to be detrimental in congestive heart failure (CHF) and that are not shared by angiotensin II. Aldosterone blockade has been associated with improved mortality in patients with left ventricular failure, already receiving an angiotensin converting enzyme inhibitor. But its role in isolated right ventricular failure has not been elucidated. The plasma arginine vasopressin levels are disproportionately elevated for the degree of serum osmolarity in patients with heart failure and result in water retention and hyponatremia. Conivaptan, a vasopressin receptor antagonist, appears to reduce body weight and improve signs of left heart failure, though there is no study to evaluate its role in right ventricular failure with edema.

This study will examine the role of spironolactone and conivaptan in patients with right ventricular failure and pathophysiology of sodium and water retention in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with World Health Organization (WHO) group 1 pulmonary arterial hypertension [51], excluding patients with portal hypertension, meeting the following hemodynamic parameters:

* Mean pulmonary artery pressure (mPAP) >35 mmHg at rest, and
* Pulmonary capillary wedge pressure (PCWP) <15 mmHg, and
* Pulmonary vascular resistance (PVR) >1.5 wood units, and 2. Age 18 to 75 years 3. Right ventricular failure defined by right atrial pressure >7 mmHg along with either dilated right ventricle, or absence of inferior vena cava collapse or BNP >100 pg/ml 4. Patients of childbearing age must be practicing effective birth control. 5. Normal left ventricular function as assessed by echocardiogram, multiple gated acquisition (MUGA) cardiac scan, or invasive left ventriculography.

Exclusion Criteria:

1. Group 2-5 pulmonary hypertension as defined by WHO.

* Pulmonary hypertension with left heart failure (as assessed by echocardiogram, multiple gated acquisition (MUGA) cardiac scan, or invasive left ventriculography).
* Pulmonary hypertension associated with lung disease and/or hypoxemia (e.g. chronic obstructive pulmonary disease, interstitial lung disease, sleep disordered breathing, chronic exposure to high altitude, alveolar hypoventilation syndrome.
* Pulmonary hypertension due to chronic thrombotic and/or embolic diseases
* Miscellaneous such as sarcoidosis, compression of pulmonary vessels by adenopathy, tumor 2. Systemic hypertension, defined as a systolic pressure >140 mmHg or a diastolic blood pressure >90 mmHg 3. Patients taking angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blockers (ARBs) 4. Pregnancy 5. Chronic kidney disease (serum creatinine > 2.5mg/dl, proteinuria >500 mg/day, hematuria) 6. Cirrhosis or portal hypertension 7. Inability to provide informed consent. 8. Allergy to conivaptan or spironolactone. 9. Active malignancy 10. Patients receiving spironolactone 11. Enrollment in other interventional studies. 12. Patients on Highly Active Antiretroviral Therapy (HAART)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cross sectional study | 18 months
  Correlation between severity of pulmonary hypertension and neurohumoral activation, Regional Blood Flow (RBF) & Transcatheter Pulmonary Valve (TPV). Acute study:electrolyte-free water and sodium excretion. Cohort Study: Composite of Cardiac index (CI),brain natriuretic peptide (BNP) and Right Atrial Pressure (RAP)

SECONDARY OUTCOMES:
Cross-sectional Study | 18 months
  Correlations between mean pulmonary artery pressure, pulmonary vascular resistance; and neurohumoral activation, glomerular filtration rate (GFR) and Transcatheter Pulmonary Valve (TPV). Acute study:correlation between response to drug and severity of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Bansal, MD, Principal Investigator — UCHSC
Locations (1):
- University of Colorado at Denver and Health Sciences Center General Clinical Research Center, Denver, Colorado, United States